CLINICAL TRIAL: NCT04089878
Title: "To Study the Impact of Balloon-occluded Retrograde Transvenous Obliteration (BRTO)/Plug Assisted Retrograde Transvenous Obliteration (PARTO) Mediated Portal Flow Modulation in Reduction of Ammonia and Improvement in Organ Volume and Functionality in Patients of Cirrhosis With LR Shunt - A Randomized Trial.ImPARTO Trial"
Brief Title: "To Study the Impact of Balloon-occluded Retrograde Transvenous Obliteration (BRTO)/Plug Assisted Retrograde Transvenous Obliteration (PARTO) Mediated Portal Flow Modulation in Reduction of Ammonia and Improvement in Organ Volume and Functionality in Patients of Cirrhosis With LR Shunt
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-25
Record Dates: First submitted 2019-08-28; First posted 2019-09-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-08

CONDITIONS: Liver Cirrhoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PARTO/BRTO + SMT (Experimental): PARTO/BRTO with SMT will be given.
  Interventions: Procedure: Plug assisted retrograde transvenous obliteration/Balloon-occluded retrograde transvenous obliteration
- Standard Medical Treatment (Active Comparator): Antibiotics, nutrition and supportive treatment
  Interventions: Other: Standard Medical Treatment

INTERVENTIONS:
Procedure: Plug assisted retrograde transvenous obliteration/Balloon-occluded retrograde transvenous obliteration — Plug assisted retrograde transvenous obliteration/Balloon-occluded retrograde transvenous obliteration
  Arms: PARTO/BRTO + SMT
Other: Standard Medical Treatment — Antibiotics, nutrition and supportive treatment
  Arms: Standard Medical Treatment

SUMMARY:
The informed consent will be obtained from the participants in the study. The study will be conducted on indoor patients, Department of Hepatology ILBS, New Delhi. This will be a Pilot study (sample size 25 cases in each arm) with 50% chances of each patient to randomized into each arm(1:1 randomization) .

Study Population - Patients with hepatic encephalopathy with LR shunt admitted in wards/HDU (High Dependency Unit)/LC ICU(Liver Coma ICU).

Study design-Randomized controlled Trial

Study period- 1 year.

Sample Size-Single Centre prospective RCT

* Sample size- Pilot study (sample size 25 cases in each arm)
* Follow up duration-6 months

ELIGIBILITY:
Inclusion Criteria:

* Child A and B cirrhotic patients with Gastro/lieno-renal shunt of >8 mm.
* Covert or Overt HE
* Age 18 to 70 years

Exclusion Criteria:

* Intractable ascites
* PVT (with 100 % block )or PV Cavernoma and splenic vein thrombosis
* High risk esophageal varices (till eradicated)
* HVPG >16 mm Hg
* HCC
* Pregnancy and lactation
* Refusal to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09-14 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in covertHepatic Encephalopathy in both groups. | 1 year
  Covert HE or overt HE will be analysed using clinical examination(west haven grading), specialised tests like stroop test, CFF(critical flicker frequency) or in rare cases EEG can be done.

SECONDARY OUTCOMES:
Change in ammonia level in both groups | 1 year
Incidence of ascites in both groups | 1 year
  Acute variceal bleed (AVB) - will be estimated by history of hematemesis, melena, and AVB will be confirm by endoscopy if these clinical history present. It can be oesophageal variceal or gastric variceal bleed as per sarin's classification, which is confirmed and managed with endoscopy procedure. AVB is defined as a bleed in a known or suspected case of PHT, with the presence of hematemesis within 24 h of presentation, and/or ongoing melena, with last melanic stool within last 24 h. The time frame for the AVB episode is 48 h. AVB is further classified as active or inactive at the time of endoscopy. BRTO/PARTO is technically feasible, safe, and effective for gastric variceal haemorrhage in patients with portal hypertension.
Incidence of acute variceal bleed in both groups. | 1 year
  Acute variceal bleed (AVB) - will be estimated by history of hematemesis, melena, and AVB will be confirm by endoscopy if these clinical history present. It can be oesophageal variceal or gastric variceal bleed as per sarin's classification, which is confirmed and managed with endoscopy procedure. AVB is defined as a bleed in a known or suspected case of PHT, with the presence of hematemesis within 24 h of presentation, and/or ongoing melena, with last melanic stool within last 24 h. The time frame for the AVB episode is 48 h. AVB is further classified as active or inactive at the time of endoscopy. BRTO/PARTO is technically feasible, safe, and effective for gastric variceal haemorrhage in patients with portal hypertension.
Number of participants with Liver transplant or death in both groups. | 1 year
Change in MELD (Model for End Stage Liver Disease) by >5 point improvement in both groups. | 6 months
  MELD: A disease severity scoring system for adults with liver disease, designed to improve the organ allocation in transplantation based on the severity of liver disease rather than the length of time on the waiting list.A MELD score is a number that ranges from 6 to 40, based on lab tests.
Change in CTP (Child-Pugh score) by 2 points improvement in both groups. | 6 months
  CTP- Child-Turcotte-Pugh score is ranges from 5 to 15, lowest is best and highest is worst .
Changes in portal flow in both groups. | 1 year
  Change will be measured by ICG and Doppler study tests.
Number of patients with prevention of Gastro-Variceal bleed in both groups. | 1 year
  It is a clinical outcome and it will be assessed by history and will be confirmed and managed by endoscopic procedure.
Number of patients with adverse effects of PARTO/BRTO (Balloon-occluded retrograde transvenous obliteration) in both groups. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dr Shiv Kumar Sarin, DM, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided